CLINICAL TRIAL: NCT04633811
Title: Effect of Weight Loss on Urinary Oxalate Excretion in Obese Calcium Oxalate Kidney Stone
Brief Title: Effect of Weight Loss on Urinary Oxalate Excretion in Obese Calcium Oxalate Kidney Stone Formers
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: University of Texas Southwestern Medical Center (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Dean Assimos, MD, Principal Investigator, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IRB-300006133; R01DK128160 (NIH)
Record Dates: First submitted 2020-11-11; First posted 2020-11-18 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Kidney Stone
MeSH Terms: conditions — Kidney Calculi

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Controlled Diet and Weight Loss Program (Experimental): Subjects will consume a low oxalate diet with blood and urine collections to establish baseline levels before undergoing a weight loss program with Optifast VLCD products. After completing the weight loss program, subjects will once again consume a low oxalate diet with blood and urine collections to observe any changes that may have occurred due to the weight loss.
  Interventions: Dietary Supplement: Low Oxalate Diet before Weight Loss; Dietary Supplement: Oral load of oxalate and sucralose before Weight Loss; Dietary Supplement: Optifast VLCD Program; Dietary Supplement: Optifast VLCD Transition Phase; Dietary Supplement: Low Oxalate Diet after Weight Loss; Dietary Supplement: Oral load of oxalate and sucralose after Weight Loss

INTERVENTIONS:
Dietary Supplement: Low Oxalate Diet before Weight Loss — Subjects will be instructed to ingest a controlled diet low in oxalate for a total of 6 days. 2 x 24 hour urines will be collected on days 3 and 4.
Dietary Supplement: Oral load of oxalate and sucralose before Weight Loss — Subjects will ingest 100mg carbon-13 oxalate, and 1 gram of sucralose on day 5 of the 6-day low oxalate diet phase. Following the oral load, blood and urine will be collected every 30 minutes and hourly, respectively
Dietary Supplement: Optifast VLCD Program — Subjects will go on a 10-week Intestive level Optifast VLCD weight loss program
Dietary Supplement: Optifast VLCD Transition Phase — After completion of the 10-week Optifast VLCD Program, subjects will be weaned off the Optifast products for 4 weeks.
Dietary Supplement: Low Oxalate Diet after Weight Loss — Subjects will be instructed to ingest a controlled diet low in oxalate for a total of 11 days and collect 2 x 24 hour urines on days 8 and 9
Dietary Supplement: Oral load of oxalate and sucralose after Weight Loss — Subjects will ingest 100mg carbon-13 oxalate, and 1 gram of sucralose on day 10 of the 11-day low oxalate diet phase. Following the oral load, blood and urine will be collected every 30 minutes and hourly, respectively

SUMMARY:
This protocol seeks to determine if weight reduction with the Optifast VLCD program leads to reduced contribution of endogenous oxalate synthesis and dietary oxalate absorption to the urinary oxalate pool in obese calcium oxalate stone formers.

DETAILED DESCRIPTION:
Obese adults (≥19 and ≤ 65 years) with a history of calcium oxalate kidney stone disease will be recruited at both University of Alabama at Birmingham (UAB) and University of Texas South Western (UTSW). Following consent, subjects will complete a screening phase, which includes (1) a meeting with a dietitian to ensure willingness to consume controlled ultra-low oxalate diets and determine anthropometric measurements and blood pressure, (2) collection of fasted blood and 2 x 24-hour urine specimens on self-choice diets to determine general health status and urinary chemistries, respectively, (3) completion of a 7-day run-in diet that includes the use of one serving of an Optifast meal daily to assess tolerance to Optifast VLCD® products. Participants will then consume an eucaloric, ultra-low oxalate controlled diet for 6 days. The controlled dietary phase involves 2 days of dietary equilibration, followed by 2 x 24-hour urine collections, and on the 5th day a dietary oxalate/sucralose oral load. Following the dietary oxalate/sucralose oral load, subjects will have blood collected every 30 minutes and collect 1-hour urines. Participants will then go on an intensive 14-week Optifast VLCD® Program to induce weight loss. At the end of this Optifast VLCD® Program participants will again perform the low oxalate controlled diet and dietary/sucralose oral load study. A total of 40 adult obese calcium oxalate kidney stone formers (20 male and 20 female) will be enrolled (20 at UAB and 20 at UTSW).

ELIGIBILITY:
Inclusion Criteria:

* First time or recurrent calcium oxalate stone formers defined as composition of most recent stone >50% calcium oxalate without uric acid component
* Last stone passage or removal greater than 3 months prior to screening
* Body Mass Index (BMI) >35 kg/m2
* Able to provide consent
* Hemoglobin A1C <6.5%
* Normal fasting blood CMP: Normal serum Na, K, Cl, CO2, Calcium, Albumin, AST, ALT <2 times upper limit of normal, Glucose <126 mg/dl, eGFR >60 ml/min/1.73 m2.
* 24-hour urine collection with creatinine within 20% of gender appropriate (mg creat/kg body weight) and consistent between collections (within 20% of each other)
* Willing to ingest menus prepared at the University of Alabama and University of Texas Southwestern Clinical Research Units
* Willing to consume the Optifast VLCD diet
* Willing to ingest menus prepared in Metabolic kitchen. No food allergies or intolerance to any of the foods in study menus. Substitutions for lactose intolerance will be made.
* Willing to avoid vigorous exercise during eucaloric, low-oxalate dietary phase
* Willing to stop use of weight-loss medications
* Willing to stop for 14 days before and during study: medications for stone prevention including diuretics, potassium citrate, allopurinol, febuxostat, and calcium, nutritional, or herbal supplements
* Those with controlled hypertension (systolic blood pressure <160 mmHg, diastolic <90 mmHg) will be included.
* Those without severe dyslipidemia (LDL <200 mg/dL, HDL >30 mg/dL, and triglycerides <250 mg/dL) will be included. Treated and controlled dyslipidemia is accepted
* Smoking/chewing tobacco/vaping will be allowed

Exclusion Criteria:

* Renal colic or past stone surgery in the past 3 months
* Estimated Glomerular Filtration Rate (eGFR) less than 60 ml/min/1.73m2
* History of type 2 diabetes or screening hgb A1c greater than or equal to 6.5%
* Alcohol or drug abuse. Alcohol consumption >12 units per week and/or unwillingness to abstain from alcohol consumption 2 days before and during the study.
* Mental/medical condition likely to impede study completion
* Current/planned pregnancy or breastfeeding in coming 6 months, unwillingness to use effective method of birth control during the study for individuals of childbearing potential.
* Planned vacation in coming 4 months
* Febrile illness including flu/common cold/COVID-19 within 21 days of study start
* Primary or enteric hyperoxaluria
* Gastrointestinal disorder or surgery that impacts oxalate transport
* Cirrhosis, pancreatic or biliary disorder, porphyria, gout
* Malignancy treated within the past 12 months
* Nephrotic syndrome, neurogenic bladder, urinary diversion
* History of primary hyperparathyroidism, cystinuria, renal tubular acidosis, sarcoidosis, cystic fibrosis
* Uncontrolled hypertension, myocardial infarction in past 6 months, unstable angina, congestive heart failure
* Medications: Topiramate, acetazolamide, zonisamide, diuretics, SGLT2-inhibitors, immunosuppressants

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2021-12-03 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Measurement of 24 hour urinary oxalate excretion | 4 days
  Subjects will ingest a controlled diet low in oxalate and collect 2 x 24-hour urines before and after the Optifast VLCD Program. The utilization of a low oxalate diet allows assessment of the change in contribution of endogenous oxalate synthesis to the urinary oxalate pool.

CONTACTS AND LOCATIONS:
Overall Officials: Dean Assimos, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No